CLINICAL TRIAL: NCT04514952
Title: Individual Patient Expanded Access IND of Autologous HBadMSCs for the Treatment of Amyotrophic Lateral Sclerosis
Status: No longer available | Type: Expanded Access
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Other Study IDs: HBALS01
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Neurodegenerative; MSCs; Stem cells; Sclerosis; ALS; Amyotrophic
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Sclerosis

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: HB-adMSCs — Hope Biosciences autologous adipose-derived mesenchymal stem cells

SUMMARY:
The drug for this submission is Hope Biosciences' autologous, adipose-derived culture-expanded mesenchymal stem cells (HB-adMSCs) for the treatment of a single patient with Amyotrophic Lateral Sclerosis (ALS). Stem cells have become a promising tool for the treatment of inflammatory and neurodegenerative conditions, including autoimmune diseases, traumatic brain injury, Parkinson's disease, and Alzheimer's disease.

DETAILED DESCRIPTION:
Once the eligibility is confirmed, approximately 1-2 weeks after the screening visit, the subject will return for the baseline/first infusion visit. Subsequent treatments will occur 2 weeks apart for 18 weeks, for a total of 10 infusions. Follow-up visits will occur at 22 weeks, 26 weeks and 39 weeks. End of study visit will occur at 52 weeks.

Baseline/Infusion 1 Visit

1. A verification of patient consent will be verbally performed and included in the progress note.
2. Review of medical history, and concomitant medications.
3. Physical exam + ALS Functional Rating Scale-Revised (ALSFRS-R)
4. Vital signs (Heart Rate, Blood Pressure, Respirations, Temp., SpO2)
5. Weight measurement
6. Blood samples will be collected for safety and efficacy assessments:

   * Hematology
   * Chemistry
   * Coagulation Panel
   * Proinflammatory Cytokines (IL-2, IL-6, TNF-a)
   * C- Reactive Protein (CRP)
7. The HB-adMSCs will be administered and the patient closely observed:

   • One intravenous infusion of HB-adMSCs (2x108 cells) to last 1 hour:

   - Saline Solution.
8. The subject will then be monitored for a minimum of 2hr after infusion as follows:

   * Measure Vital signs at minute 0 of infusion.
   * Measure Vital signs at minute 15 after IV infusion.
   * Measure Vital Signs at minute 30 after IV infusion.
   * Measure Vital signs at minute 60 after IV infusion.
   * Measure Vital signs at minute 120 after IV infusion. (Vital signs will be recorded more frequently if clinically indicated).
9. Adverse event monitoring
10. 24 hrs. Telephone encounter. The subject will be contacted by telephone the following day after the infusion visit to determine if any adverse events have occurred.
11. ALS-specific Quality of Life Survey-revised (ALSSQOL-R)
12. A video recording will be made with the purpose to capture patient's overall status (gait, range of motion assessments, etc.).

One week following infusion, PI will perform an assessment to determine patient status and discuss any changes since previous infusion.

Infusion Visits Week 2,6,10,14 and 18

1. Review and update medical history
2. Update concomitant medications list
3. Weight measurement
4. Vital signs (Heart Rate, Blood Pressure, Respirations, Temp., SpO2)
5. Physical examination + ALS Functional Rating Scale-Revised (ALSFRS-R)
6. The HB-adMSCs will be administered and the patient closely observed:

   • One intravenous infusion of HB-adMSCs (2x108 cells) to last 1 hour:

   - Saline Solution.
7. Adverse event monitoring
8. 24 hrs. Telephone encounter. The subject will be contacted by telephone the following day after the infusion visit to determine if any adverse events have occurred.

Infusion Visits Week 4, 8, 12, and 16

1. Review and update medical history
2. Update concomitant medications list
3. Weight measurement
4. Vital signs (Heart Rate, Blood Pressure, Respirations, Temp., SpO2)
5. Physical examination and ALS Functional Rating Scale-Revised (ALSFRS-R)
6. Blood samples will be collected for safety and efficacy assessments:

   * Hematology
   * Chemistry
   * Coagulation Panel
   * Proinflammatory Cytokines (IL-2, IL-6, TNF-a)
   * C - Reactive Protein
7. The HB-adMSCs will be administered and the patient closely observed:

   • One intravenous infusion of HB-adMSCs (2x108 cells) to last 1 hour:

   - Saline Solution.
8. ALS-specific Quality of Life Survey-revised (ALSSQOL-R)
9. Adverse event monitoring
10. 24 hrs. Telephone encounter. The subject will be contacted by telephone the following day after the infusion visit to determine if any adverse events have occurred.

Follow-Up Visit Week 22

1. You will be asked about your current health and medical history (if any changes since last study visit or telephone call).
2. You will be asked if there was any change in the medication list you have previously provided (Concomitant medication list).
3. Your blood pressure, heart rate, respiration rate, temperature, oxygen saturation and weight will be measured.
4. The doctor will perform a physical examination driven by the signs and/or symptoms you experience, if any.
5. The doctor will perform tests including the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) to measure the symptoms of ALS Disease on how you are able to perform.
6. You will be asked to complete the Amyotrophic Lateral Sclerosis-Specific Quality of Life-Revised (ALSSQOL-R) questionnaire to assess the impact of Amyotrophic Lateral Sclerosis on your quality of life.
7. You will be reminded to stay on your stable regimen of treatment throughout the study

Follow-Up Visit Week 26

1. You will be asked about your current health and medical history.
2. You will be asked about the medicines that you have taken and are currently taking for Amyotrophic Lateral Sclerosis and for other health issues.
3. Your blood pressure, heart rate, respiration rate, oxygen saturation, temperature, and weight will be measured.
4. The doctor will perform a complete physical examination.
5. The doctor will perform tests including the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) to measure the symptoms of ALS Disease on how you are able to perform.
6. You will be asked to complete the Amyotrophic Lateral Sclerosis-Specific Quality of Life-Revised (ALSSQOL-R) questionnaire to assess the impact of Amyotrophic Lateral Sclerosis on your quality of life.
7. Laboratory test will be done. Your blood will be tested to measure your overall health and efficacy markers (TNF-a, IL-6, IL-2 and C - Reactive Protein).
8. You will be given an order for a Chest X ray (PA single view) and Magnetic Resonance Imaging to be performed. If within 7 days of the End of study visit you have undergone any or both, such reports would suffice this requirement.
9. An Electrocardiogram (ECG) will be performed to evaluate cardiac function.
10. An Electromyogram (EMG) will be performed to evaluate neuromuscular function.
11. A video documenting of yourself walking and sitting will be performed.

Follow-Up Visit Week 39

1. You will be asked about your current health and medical history (if any changes since last study visit or telephone call).
2. You will be asked if there was any change in the medication list you have previously provided (Concomitant medication list).
3. Your blood pressure, heart rate, respiration rate, temperature, oxygen saturation and weight will be measured.
4. The doctor will perform a physical examination driven by the signs and/or symptoms you experience, if any.
5. Laboratory test will be done. Your blood will be tested to measure your overall health and efficacy markers (TNF-a, IL-6, IL-2 and C - Reactive Protein).
6. The doctor will perform tests including the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) to measure the symptoms of ALS Disease on how you are able to perform.
7. You will be asked to complete the Amyotrophic Lateral Sclerosis-Specific Quality of Life-Revised (ALSSQOL-R) questionnaire to assess the impact of Amyotrophic Lateral Sclerosis on your quality of life.
8. You will be reminded to stay on your stable regimen of treatment throughout the study

End of Study Visit Week 52

1. Review and update medical history
2. Review and update concomitant medications list
3. Weight measurement
4. Vital signs (Heart Rate, Blood Pressure, Respirations, Temp., SpO2)
5. Physical examination + ALS Functional Rating Scale-Revised (ALSFRS-R)
6. Blood samples will be collected for safety and efficacy assessments:

   * Hematology
   * Coagulation Panel
   * Proinflammatory Cytokines (IL-2, IL-6, TNF-a)
   * C - Reactive Protein
7. ALS-specific Quality of Life Survey-revised (ALSSQOL-R)
8. Chest X-Ray (PA single view)
9. Electromyogram (EMG)
10. Magnetic Resonance Imaging (MRI)
11. Adverse event monitoring
12. A video recording will be made with the purpose to capture patient's overall status (gait, range of motion assessments, etc.).

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of Amyotrophic Lateral Sclerosis.
2. Capable of giving informed consent (signed, verbal or assent as applicable and as listed in the protocol)

Exclusion Criteria:

1. Other acute or chronic medical conditions that, in the opinion of the investigator, may increase the risks associated with study participation or HB-adMSCs administration.
2. Any abnormal, inexplicable laboratory result that, in the opinion of the investigator, may increase the risks associated with study participation or HB-adMSCs administration.
3. Participation in other interventional research studies within the past 30 days.
4. Unwillingness to return for follow-up visits.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Thakur, MD, Principal Investigator — River Oaks Hospital and Clinics
Locations (1):
- River Oaks Hospital and Clinics, Houston, Texas, United States